CLINICAL TRIAL: NCT01538121
Title: Antiphospholipid Antibodies and Early Severe Preeclampsia (< 34 Weeks of Gestation). A Case-Control Study.
Brief Title: Antiphospholipid Antibodies and Early Severe Preeclampsia.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., MD, Saint Thomas Hospital, Panama
Other Study IDs: MHST2012-01A
Record Dates: First submitted 2012-02-19; First posted 2012-02-23 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Severe Preeclampsia; Antiphospholipid Syndrome
Keywords: Antibodies, anticardiolipin; Antibodies, B2 Glycoprotein I; Lupus Anticoagulant; Severe Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia; Antiphospholipid Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases-Early Severe Preeclampsia: Patients with severe preeclampsia before 34 weeks of gestation
- Controls: Patients with normal pregnancies at term.

SUMMARY:
The Antiphospholipid Syndrome is an immune disease where the presence of antibodies directed against cell membrane phospholipids (antiphospholipid antibodies) can cause an hypercoagulable state that causes thrombosis and obstetric complications (miscarriages, stillbirths). Since 1999 the Sapporo Criteria for Antiphospholipid Syndrome diagnosis includes the development of severe preeclampsia before 34 weeks of gestation, but this was done without solid evidence of a relation between the two. Our study will try to add information to this particular point.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 24-34 weeks
* Diagnosis of severe preeclampsia

Exclusion Criteria:

* Known antiphospholipid syndrome.
* Known presence of antiphospholipid antibodies.
* Patients with systemic lupus erythematosus.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant patients admitted for severe preeclampsia between 24-34 weeks pf gestation (cases) and normal patients in labor at term (controls).
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Lupus anticoagulant | 15 months
  Number of cases positive for Lupus Anticoagulant.
Anticardiolipin antibodies | 15 months
  Number of cases with high/medium levels of IgG/IgM of anticardiolipin antibodies.
B2 Glycoprotein I | 15 months
  Number of cases with levels of B2 Glycoprotein 1 > 99%

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo A Reyes, MD, Principal Investigator — Saint Thomas Hospital, Panama
Locations (1):
- Saint Thomas Maternity Hospital, Panama City, Provincia de Panamá, Panama